CLINICAL TRIAL: NCT01411852
Title: Field Trial of Hypotensive Resuscitation Versus Standard Resuscitation in Patients With Hemorrhagic Shock After Trauma: A Pilot Trial
Brief Title: Field Trial of Hypotensive Versus Standard Resuscitation for Hemorrhagic Shock After Trauma
Acronym: HypoResus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Susanne May, PhD/Principal Investigator, Resuscitation Outcomes Consortium Data Coordinating Center, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41071-B; 5U01HL077863-07 (NIH)
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Blunt Trauma; Penetrating Wound; Hemorrhagic Shock
Keywords: fluid volume resuscitation; trauma; hemorrhagic shock
MeSH Terms: conditions — Wounds, Nonpenetrating; Wounds, Penetrating; Shock, Hemorrhagic; Wounds and Injuries | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.9% Sodium Chloride 250 mL bolus (Experimental): 0.9% Sodium Chloride 250 mL bolus - A large bore IV will be placed and a 250cc bag of normal saline (NS) will be hung. If IV placement is difficult, NS can be given through an intraosseous line. Using small bags versus large bags will physically limit the amount of fluid given to patients in the experimental group. The requirement to change the smaller bags of fluid and recheck the pulse or blood pressure will limit the amount of fluid given. The procedure will continue until 2 hours after arrival to the hospital or until hemorrhage control is achieved whichever occurs first. Hemorrhage control will be defined as ligation of a bleeding vessel, packing of a solid organ, removal of a solid organ, and angiographic embolization of a bleeding vessel.
  Interventions: Drug: 0.9% Sodium Chloride 250 mL bolus
- 0.9% Sodium Chloride 2000 mL bolus (Active Comparator): 0.9% Sodium Chloride 2000 mL bolus - The treatment of the control group will be consistent with traditional Prehospital Trauma Life Support and Advanced Trauma Life Support guidelines which recommend early aggressive fluid resuscitation. An intravenous line (IV) will be placed and a 1000cc bag of normal saline will be hung. If IV placement is difficult, fluid can be given through an intraosseous line. This procedure will continue until either 2 hours after hospital arrival or until control of hemorrhage is achieved whichever occurs first. Hemorrhage control will be defined as ligation of a bleeding vessel, packing of a solid organ, removal of a solid organ, and angiographic embolization of a bleeding vessel.
  Interventions: Drug: 0.9% Sodium Chloride 2000 mL bolus

INTERVENTIONS:
Drug: 0.9% Sodium Chloride 250 mL bolus — Emergency Medicine Systems (EMS) agencies and in-hospital providers will be given the option to utilize either systolic blood pressure (SBP) or radial pulse as the endpoint for fluid resuscitation to patients randomized to the experimental group. Patients will receive a 250 ml bolus of normal saline (NS) only if the SBP is less than 70 mmHg or the radial pulse is not palpable. If the SBP is greater than or equal to 70 mmHg or the radial pulse is palpable, NS will be given to keep the vein open. The presence or absence of a radial pulse or the SBP will be documented before and after each bolus. The study will continue repeating the randomization procedure using only 250 ml bags of NS until 2 hours after arrival to the hospital or until hemorrhage control is achieved whichever occurs first.
  Other Names: isotonic saline; normal saline
  Arms: 0.9% Sodium Chloride 250 mL bolus
Drug: 0.9% Sodium Chloride 2000 mL bolus — Emergency Medicine Systems (EMS) personnel and in-hospital providers will utilize the systolic blood pressure SBP as the endpoint for delivering fluid resuscitation to patients randomized to the control group. If the SBP is equal to or less than 90 mmHg, the EMS personnel will start infusing a 1000 ml bolus of normal saline (NS) and will continue using only 1000 ml bags of NS as needed. If the total fluid resuscitation exceeds 2 liters, fluid will be stopped when the SBP exceeds 110 mmHg and restarted as necessary to maintain a goal SBP of 110 mmHg. The fluid will be given as rapidly as possible. This fluid resuscitation protocol will continue until either 2 hours after hospital arrival or until control of hemorrhage is achieved whichever occurs first.
  Other Names: isotonic saline; normal saline
  Arms: 0.9% Sodium Chloride 2000 mL bolus

SUMMARY:
Primary Aim: To determine the feasibility and safety of hypotensive resuscitation for the early treatment of patients with traumatic shock compared to standard fluid resuscitation.

Primary Hypotheses: The null hypothesis regarding feasibility is that hypotensive resuscitation will result in the same volume of early crystalloid (normal saline) fluid administration compared to standard crystalloid resuscitation. The null hypothesis regarding safety is that hypotensive resuscitation will result in the same percent of patients surviving to 24 hours after 911 call received at dispatch compared to standard fluid resuscitation. Early resuscitation is defined as all fluid given until 2 hours after arrival in the Emergency Department or until hemorrhage control is achieved in the hospital, whichever occurs earlier.

DETAILED DESCRIPTION:
1. Overview This multi-center pilot trial is designed to determine the feasibility and safety of hypotensive resuscitation for the early resuscitation of patients with traumatic shock compared to standard fluid resuscitation. Blunt and penetrating trauma patients with a prehospital systolic blood pressure (SBP) ≤ 90 mmHg will be eligible. In the hypotensive resuscitation group, an intravenous line (IV) will be placed and a radial pulse will be palpated. If the radial pulse is present or the SBP is greater than or equal to 70, a 250 ml bag of normal saline will be hung and maintained at a keep the vein open rate only. If the radial pulse is absent, the 250 ml of normal saline will be given as a bolus. This process using small bags of fluid will be repeated until a radial pulse is palpable or until 2 hours after Emergency Department (ED) arrival or until hemorrhage control has been achieved. The decision to utilize a SBP versus a radial pulse will be made a priori. Patients in the standard fluid resuscitation group will have an IV placed and a 1000 ml bag of normal saline (NS) will be hung. Fluid will be given as rapidly as possible and continued until hospital arrival. If the prehospital or hospital fluid resuscitation exceeds 2 liters, it will be stopped when the SBP exceeds 110 mmHg and restarted as necessary to maintain a goal SBP of 110 mmHg. This randomization scheme will be continued for 2 hours after hospital arrival or until hemorrhage control is achieved whichever occurs first. The randomization will not affect the indications for the administration of blood products but we hypothesize that less blood products and total fluid will be given in the experimental group due to avoidance of the pop-the-clot phenomenon, less hemodilution and less coagulopathy.

   Patients who experience ground level falls are characterized as having low injury severity scores. (70) Patients with suspected ground level falls will be excluded in an effort to focus enrollment on the more severely injured patients at risk for trauma related hemorrhagic shock. Patients with severe traumatic brain injury will be excluded due to lack of equipoise. In observational studies (1-5) a relationship between hypotension and poor neurologic outcomes has been observed and EMS personnel as well as researchers at this time believe that it is unethical to withhold resuscitation fluid from patients with traumatic brain injury. Patients with suspected spinal cord injury will also be excluded based on evidence that indicates they are at risk for cardiovascular failure due to hemodynamic compromise correlated with the presence of neurogenic hypotension at the time of hospital admission. (69) All enrolled patients will be retrospectively screened to determine if they had evidence of severe traumatic brain injury with GCS≤8 or spinal cord injury at the time of enrollment.

   Screening information will be obtained for all potentially eligible patients who meet all inclusion criteria. Screening will also document whether each exclusion criterion is met. The rate at which screened patients were enrolled and later found to have met one or more of the exclusion criteria will be assessed to determine if the inclusion and exclusion criteria need to be adjusted to avoid enrollment of these patients for future studies. These patients will also be assessed to determine if enrollment in the protocol potentially harmed these patients.

   The study will be a two arm, randomized interventional trial comparing the two resuscitation strategies. Due to obvious differences in the treatment of enrolled patients, the study will not be blinded. Nevertheless, treatment bags will be packaged in containers such that providers will not be able to identify whether treatment containers house 1000 ml bags or 250 ml bags until the treatment containers are opened. The patient will be considered randomized at the time a study bag is opened regardless of whether any fluid is given or not. Hospitals will be provided with 250 ml bags of NS to continue treatment of those patients randomized to the hypotensive resuscitation arm.

   The primary outcomes of the study will be volume of prehospital and in-hospital fluid administered from time of injury until 2 hours into the hospital stay or until hemorrhage is controlled to test feasibility and 24 hour survival for the safety hypothesis. Secondary outcomes will include measures of protocol adherence, 24 hour fluid volume, 24 hour blood product requirements, ventilator days, hospital length of stay, intensive care unit (ICU) length of stay, admission base deficit, development of renal failure, admission hematocrit and admission coagulation parameters. The primary goals of this pilot study will be to determine if the described model will result in different early fluid volumes being delivered to the two groups and to determine if these differing volumes impact mortality. If this pilot study shows that hypotensive resuscitation is feasible and safe, a larger trial will be planned to determine the efficacy of hypotensive fluid resuscitation.

   This study will be conducted by the Resuscitation Outcomes Consortium (ROC) which is a collaboration of 7 regional sites in the United States and Canada and a Data Coordinating Center. This consortium is charged with the task of conducting clinical trials in patients with life threatening trauma and cardiac arrest. The following ROC sites have committed to participating in this trial: Alabama, Dallas, Milwaukee, Ottawa, Pittsburgh, Portland, and Vancouver.
2. Specific Aims and Hypotheses Specific Aim 1: To investigate whether early crystalloid (normal saline) resuscitation volume can be reduced for trauma patients with hemorrhagic shock who receive hypotensive resuscitation versus those who receive standard early resuscitation (feasibility) and whether there are differences in 24-hour survival between the groups (safety).

Primary Hypotheses: The null hypothesis is that patients who receive hypotensive resuscitation and patients who receive standard resuscitation will have the same volume of early crystalloid (normal saline) resuscitation administered and will have the same 24-hour survival from 911 call received at dispatch time.

Specific Aim 2: To assess protocol adherence and differences in morbidity and adverse events for hypotensive versus standard resuscitation.

Secondary Hypotheses: The null hypotheses are that protocol adherence is low and that hypotensive resuscitation versus standard resuscitation will result in the same amount of total fluid volume and total blood product requirements within 24 hours from 911 call received at dispatch, the same base deficit, hematocrit and coagulation parameters on admission to the ED, number of days on a ventilator, duration of hospital stay, ICU length of stay, and incidence of renal failure.

ELIGIBILITY:
Inclusion Criteria: Included will be those with:

* Blunt or penetrating injury
* Age ≥15yrs or weight ≥50kg if age is unknown
* Prehospital SBP ≤ 90 mmHg

Exclusion Criteria: Excluded will be those with:

* Ground level falls
* Evidence of severe blunt or penetrating head injury with a Glasgow Coma Scale (GCS) ≤ 8
* Bilateral paralysis secondary to suspected spinal cord injury
* Fluid greater than 250ml was given prior to randomization
* Cardiopulmonary resuscitation (CPR) by Emergency Medicine Service (EMS) prior to randomization
* Known prisoners
* Known or suspected pregnancy
* Drowning or asphyxia due to hanging
* Burns over a Total Body Surface Area (TBSA) > 20%
* Time of call received at dispatch to study intervention > 4 hours

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron L Weisfeldt, MD, Study Chair — Resuscitation Outcomes Consortium; David Hoyt, MD, Study Director — Resuscitation Outcomes Consortium
Locations (6):
- United States (5):
  - Alabama Resuscitation Center, University of Alabama, Birmingham, Alabama
  - Portland Resuscitation Outcomes Consortium, Oregon Health & Sciences University, Portland, Oregon
  - The Pittsburgh Resuscitation Network, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Dallas Center for Resuscitation Research, University of Texas Southwestern Medical Center, Dallas, Texas
  - Milwaukee Resuscitation Network, Medical College of Wisconsin, Milwaukee, Wisconsin
- Resuscitation Outcomes Consortium Regional Coordinating Center,University of British Columbia, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled and randomized in the out-of-hospital setting. Nineteen Emergency Medical Service (EMS) systems and 10 hospital in 6 regions of the Resuscitation Outcomes Consortium (ROC) participated.
Groups:
- 0.9% Sodium Chloride 2000 mL Bolus: 0.9% Sodium Chloride 2000 mL bolus - An intravenous line (IV) will be placed and a 1000cc bag of normal saline will be hung. If IV placement is difficult, fluid can be given through an intraosseous line. This procedure will continue until either 2 hours after hospital arrival or until control of hemorrhage is achieved whichever occurs first.
  0.9% Sodium Chloride 2000 mL bolus: The systolic blood pressure (SBP) is the endpoint for delivering fluid resuscitation to patients randomized to the control group. If the SBP is equal to or less than 90 mmHg, the EMS personnel will start infusing a 1000 ml bolus of normal saline (NS) and will continue using only 1000 ml bags of NS as needed. Once the total fluid reaches 2 liters and the SBP exceeds 110 mmHg, the fluid will be stopped and restarted as necessary to maintain a goal SBP of 110 mmHg.
- 0.9% Sodium Chloride 250 mL Bolus: 0.9% Sodium Chloride 250 mL bolus - A large bore IV will be placed and a 250cc bag of normal saline (NS) will be hung. If IV placement is difficult, NS can be given through an intraosseous line. The procedure will continue until 2 hours after arrival to the hospital or until hemorrhage control is achieved whichever occurs first.
  0.9% Sodium Chloride 250 mL bolus: Either systolic blood pressure (SBP) or radial pulse is the endpoint for fluid resuscitation to patients randomized to the experimental group. Patients receive 250 ml bolus of normal saline (NS) only if the SBP is less than 70 mmHg or the radial pulse is not palpable. If the SBP is greater than or equal to 70 mmHg or the radial pulse is palpable, NS is given only to keep the vein open. The study will continue repeating the randomization procedure using only 250 ml bags of NS until 2 hours after arrival to the hospital or until hemorrhage control is achieved whichever occurs first.
Period: Prehospital Intervention Phase
Arm/Group | 0.9% Sodium Chloride 2000 mL Bolus | 0.9% Sodium Chloride 250 mL Bolus
Started | 95 (1 patient randomized to 2000 mL bolus arm but received 250 mL bolus. Analyzed in 2000 mL arm.) | 96 (One patient was in police custody at the time of enrollment. Patient's data omitted from analyses.)
Completed | 83 (12 patients had the intervention stopped prior to hospital arrival) | 89 (7 patients had intervention stopped prior to hospital arrival)
Not Completed | 12 | 7
Not completed — No qualifying SBP | 5 | 4
Not completed — Cardiopulmonary resuscitation (CPR) | 2 | 2
Not completed — Found to be under age | 0 | 1
Not completed — Severe head injury with GCS≤8 | 5 | 0
Period: Hospital Intervention Phase
Arm/Group | 0.9% Sodium Chloride 2000 mL Bolus | 0.9% Sodium Chloride 250 mL Bolus
Started | 83 | 89
Completed | 59 (24 patients had intervention stopped prior to 2 hours after arrival or hemorrhage control) | 71 (18 patients had intervention stopped prior to 2 hours after arrival or hemorrhage control)
Not Completed | 24 | 18
Not completed — Severe head injury | 5 | 4
Not completed — No qualifying SBP | 5 | 1
Not completed — Miscommunication error | 1 | 2
Not completed — CPR administered | 3 | 1
Not completed — Misunderstanding of protocol | 4 | 1
Not completed — Diagnosis of sepsis | 0 | 2
Not completed — Diagnosis of dehydration | 0 | 1
Not completed — Physician/hospital staff noncompliance | 0 | 4
Not completed — Other ineligible | 2 | 2
Not completed — Spinal cord injury | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Vascular access failed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic, Injury, and Out-of-Hospital Care Characteristics
Groups:
- Standard Resuscitation (SR): Patients in the SR group received 2 liters of fluid as an initial bolus. Following the initial bolus, additional fluid was given a needed to maintain a SBP of 110 mmHg for the duration of the study period.
- Controlled Resuscitation (CR): Patients in the CR group received a 250 milliliter (ml) bolus of saline only if their SBP was < 70 millimeters of mercury (mmHg) or they had no palpable radial pulse.
- Total: Total of all reporting groups
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR) | Total
Number analyzed (Participants) | 95 | 96 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (19.2) | 41.9 (20.2) | 41.8 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 74 | 72 | 146
Penetrating trauma [Number; unit: participants]
  Penetrating primary mechanism of injury | 33 | 32 | 65
  Blunt force primary mechanism of injury | 62 | 63 | 125
  Neither penetrating or blunt force | 0 | 1 | 1
Injury Severity Score (ISS) [Median (Inter-Quartile Range); unit: units on a scale] — The ISS is an anatomical scoring system that provides an overall score for patients with multiple injuries. Each injury is assigned an Abbreviated Injury Scale (AIS) score and is allocated to one of six body regions (Head, Face, Chest, Abdomen, Extremities (including Pelvis), External). The highest AIS score in each body region is used. The 3 most severely injured body regions have their score squared and added together to produce the ISS score. The ISS score takes values from 0 to 75. If an injury is assigned an AIS of 6 (unsurvivable injury), the ISS score is automatically assigned to 75.
  units on a scale | 9 [2 to 24.2] | 9.5 [1.8 to 19.2] | 9 [2 to 20]
Injury Severity Score (ISS): Number of Severely Injured [Number; unit: participants] — An ISS > 15 is considered severely injured. One patient died prior to hospital arrival and could not be scored.
  The ISS is an anatomical scoring system with values from 0 to 75. Each injury is assigned an Abbreviated Injury Scale (AIS) score and is allocated to one of six body regions (Head, Face, Chest, Abdomen, Extremities (including Pelvis), External). Only the highest AIS score in each region is used. The 3 most severely injured body regions have their score squared and added together to produce the ISS score. If an AIS is 6 (unsurvivable injury), the ISS is automatically scored as 75.
  participants
    Severely injured with ISS > 15 | 32 | 33 | 65
    Mildly injured with ISS ≤ 15 | 62 | 63 | 125
    Died in field with no AIS available | 1 | 0 | 1
Glasgow Coma Score (GCS) prior to enrollment [Mean (Standard Deviation); unit: units on a scale] — GCS is a reliable, objective way of recording the conscious state of a person. A patient is given a score between 3 (deep unconsciousness) and 15 (opens eyes spontaneously, alert & oriented, and obeys commands).
  Eye: 1 - no eye opening; 2 - eye opening to pain stimulus; 3 - eye opening to speech; 4 - eye opening spontaneously
  Verbal: 1 - no verbal; 2 - incomprehensible sounds; 3 - inappropriate words; 4 - confused; 5 - oriented
  Motor: 1 - no moving; 2 - decerebrate posture; 3 - decorticate posture; 4 - withdraws from pain; 5 - localizes to pain; 6 - obeys commands
  units on a scale | 12.4 (4.1) | 13 (3.6) | 12.7 (3.9)
Advanced airway [Number; unit: participants] — Insertion of an advanced airway by paramedics prior to hospital arrival
  participants
    Number of patients with advanced airway inserted | 12 | 7 | 19
    Number of patients with no advanced airway | 83 | 89 | 172
Revised Trauma Score (RTS) [Mean (Standard Deviation); unit: units on a scale] — The first GCS, SBP and Respiratory Rate (RR) are coded 4 to 0.
  4 = GCS 13-15, SBP>89, RR 10-29; 3 = GCS 9-12, SBP 26-89, RR>29; 2 = GCS 6-8, SBP 50-75, RR 6-9;
  1 = GCS 4-5, SBP 1-49, RR 1-5; 0 = GCS 3, SBP 0, RR 0
  Enter GCS, SBP, RR codes:
  RTS = 0.9368 GCS + 0.7326 SBP + 0.2908 RR
  The RTS range is 0 to 7.8408. The RTS is heavily weighted towards the GCS to compensate for major head injury without multisystem injury or major physiological changes. A threshold of RTS < 4 has been proposed to identify those patients who are severely injured and should be treated in a trauma center.
  units on a scale | 6.4 (1.7) | 6.5 (1.4) | 6.5 (1.6)
Initial SBP [Median (Inter-Quartile Range); unit: mmHg] — Time of first recorded SBP by paramedic upon arrival at injured patient's side
  mmHg | 84 [74.5 to 94] | 81.5 [72 to 92] | 84 [72 to 93]
Qualifying SBP [Median (Inter-Quartile Range); unit: mmHg] | 82 [72 to 89] | 78 [69.8 to 85] | 80 [70 to 87]
Initial heart rate (HR) [Mean (Standard Deviation); unit: number of heart beats per minute] | 91.9 (24.2) | 94.7 (22.9) | 93.3 (23.5)
Air transport [Number; unit: participants] — Number of patients who required air transport by helicopter accompanied by paramedic, registered nurse or physician. Criteria for transporting the patient by air include severity of injury and geographical barriers to transport by ground vehicle
  participants
    Number transported by air | 6 | 5 | 11
    Number transported by ground | 88 | 91 | 179
    Number died prior to transport | 1 | 0 | 1
Time from dispatch call to first intravenous/intraosseous access (IV/IO) [Mean (Standard Deviation); unit: minutes] — Number of minutes from time of call to dispatch to the recorded time of the first successful intravenous catheter (IV) insertion and intraosseous needle (IO) insertion
  minutes | 22.1 (9.9) | 21 (8.7) | 21.5 (9.3)
Total out-of-hospital time [Mean (Standard Deviation); unit: minutes] — Total number of minutes from estimated time of injury to time of hospital arrival
  minutes | 41 (13.8) | 42.7 (16.5) | 41.9 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Total Volume of All Crystalloid Given for Early Resuscitation (Feasibility)
Description: The primary feasibility endpoint was early crystalloid volume (ECV) defined as crystalloid infused from Emergency Medical Services (EMS) arrival at the scene until the end of the study period
Time Frame: From time of first intravenous or intraosseous insertion through the first 2 hours after hospital arrival or hemorrhage control, which ever occurs first
Population: Patients with traumatic shock due to blunt or penetrating mechanisms
Measure: Mean (95% Confidence Interval); unit: liters
Groups:
- ECV Difference [Standard - Controlled]: ECV treatment difference between SR and CR
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR) | ECV Difference [Standard - Controlled]
Number analyzed (Participants) | 95 | 96 | 191
liters | 2.04 [1.76 to 2.32] | 1.04 [0.75 to 1.34] | 1 [0.6 to 1.4]

2. Primary Outcome: 24 Hour Mortality
Description: The 24 hour mortality endpoint for the total number of patients each arm
Time Frame: From time of hospital arrival through the first 24 hours
Population: All patients except for one who was enrolled while in police custody
Measure: Number; unit: participants
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 95 | 96
participants
  Died within first 24 hours after hospital arrival | 14 | 5
  Alive at 24 hours after hospital arrival | 81 | 91
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.12 to 1.25] — Adjusted for age (linear spline with knot at 45 years), penetrating vs. blunt or no trauma (1 patient had neither blunt nor penetrating trauma), and Injury Severity Score (ISS). ISS multiply imputed for one patient

3. Secondary Outcome: Number of Ineligible Patients Enrolled at the Time of Randomization
Description: Eligibility criteria:
  Inclusion Criteria
  Included will be those with:
  1. Blunt or penetrating injury
  2. Age ≥15yrs or weight ≥50kg if age is unknown
  3. Prehospital SBP ≤ 90 mmHg 5.3 Exclusion Criteria
  Excluded will be those with:
  1. Ground level falls
  2. Evidence of severe blunt or penetrating head injury with a Glasgow Coma Score (GCS) ≤ 8
  3. Bilateral paralysis secondary to suspected spinal cord injury
  4. Fluid greater than 250 ml was given prior to randomization
  5. Cardiopulmonary resuscitation (CPR) by Emergency Medical Services (EMS) prior to randomization
  6. Known prisoners
  7. Known or suspected pregnancy
  8. Drowning or asphyxia due to hanging
  9. Burns Total Body Surface Area (TBSA) > 20%
  10. Time of call received at dispatch to study intervention > 4 hours
Time Frame: From the time the paramedic with study drug kit arrived at patient's side to the time kit was opened prior to ED arrival
Population: All patients enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 95 | 97
participants | 24 | 9
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; percent difference = -16.0, 95% CI 2-sided [-26.5 to -5.5]

4. Secondary Outcome: Total Fluid Requirement During First 24 Hours
Description: Total volume of fluid administered during the first 24 hours inclusive of crystalloids, blood products, 3% saline, mannitol, and other colloids
Time Frame: From ED arrival through the first 24 hours
Population: All patients except one who was enrolled while in police custody
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 95 | 96
Liters | 4.43 (4.02) | 5.61 (6.71)
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-2.76 to 0.40]

5. Secondary Outcome: Total Blood Product Requirements in First 24 Hours
Description: Total amount of blood products required: packed red blood cells (PRBC), fresh frozen plasma (FFP), platelets (plts), cryoprecipitate (cryo)
Time Frame: From ED arrival through the first 24 hours
Population: All patients except one who was enrolled while in police custody
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 95 | 96
Liters | 0.84 (2.24) | 1.61 (3.53)
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.61 to 0.08]

6. Secondary Outcome: Base Deficit on Admission to the Emergency Department (ED)
Description: The first base deficit value reported from arterial blood lab work drawn after arrival in the final Emergency Department. This measure reflects the acid-base balance in the arterial blood. A negative number indicates that the blood is more acid that normal.
Time Frame: From final Emergency Department arrival time through first 24 hours
Population: Patient with the first base deficit recorded in the first 24 hours of the ED arrival
Measure: Mean (Standard Deviation); unit: mmol/Liter
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 55 | 58
mmol/Liter | 6.4 (5.2) | 6.2 (5.7)
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.8 to 2.2]

7. Secondary Outcome: Hemoglobin on Admission to the Emergency Department
Description: The first hemoglobin value reported from blood drawn in the final Emergency Department
Time Frame: From final Emergency Department arrival time through first 24 hours
Population: All patients with a first hemoglobin measured within the first 24 hours of ED arrival
Measure: Mean (Standard Deviation); unit: grams/deciliter
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 86 | 89
grams/deciliter | 12.6 (2.1) | 12.3 (2.3)
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.3 to 1.0]

8. Secondary Outcome: Platelet Value on Admission
Description: First platelet value from blood drawn in the the first 24 hours after arrival
Time Frame: From final Emergency Department arrival time through first 24 hours
Population: All patients with the first platelet value measured within the first 24 hours of ED arrival
Measure: Mean (Standard Deviation); unit: 10^9 Platelets/Liters
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 83 | 86
10^9 Platelets/Liters | 219.5 (61.8) | 239.9 (82.4)
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Mean Difference (Final Values) = -20.4, 95% CI 2-sided [-42.5 to 1.6]

9. Secondary Outcome: International Normalized Ratio (INR) on Admission to the Emergency Department
Description: The first International normalized ratio (INR) value reported from blood drawn within the first 24 hours from arrival
Time Frame: From final Emergency Department arrival time through first 24 hours
Population: Patients who had a first INR value measured within the first 24 hours of ED arrival
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 74 | 74
ratio | 1.18 (0.26) | 1.16 (0.25)
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.06 to 0.10]

10. Secondary Outcome: Hemorrhage Control Procedure Within 2 Hours of ED Arrival
Description: Hemorrhage control procedures include blood vessel ligated or embolized, organ packed or removed, laparotomy or thoracotomy
Time Frame: From ED arrival through the first 2 hours
Population: All patients except for 1 patient who was enrolled while in police custody
Measure: Number; unit: participants
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 95 | 96
participants | 19 | 29
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; percent difference = -10.2, 95% CI 2-sided [-22.4 to 2.0]

11. Secondary Outcome: Acute Renal Failure Classification Score of "Risk" Without Glomerular Filtration Rate (GFR)
Description: Increased plasma creatinine > 1.5 x reference measure (ED admission). Urine criteria is based on 6-hour periods for this level of the RIFLE and cannot be assessed since study data are collected for 24-hour periods. This row includes patients who met the "Injury" and "Failure" criteria as well. Only measured for patients with at least 2 days of ICU stay assessed.
Time Frame: From ED arrival through Day 28
Population: Patients with at least a 2 day ICU stay
Measure: Number; unit: participants
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 24 | 35
participants | 3 | 11
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; percent difference = -18.9, 95% CI 2-sided [-39.2 to 1.4]

12. Secondary Outcome: Acute Renal Failure Classification Score of "Injury" Without Glomerular Filtration Rate (GFR)
Description: Increased plasma creatinine > 2 x reference measure (ED admission) or urine output < 0.5 mL/kg/h x 24h. The RIFLE urine criterion for this level actually specifies a 12 hour period of assessment but study data are collected for 24-hr periods. This row includes patients who met the "Failure" criteria as well. Only measured for patients with at least 2 days of ICU stay assessed.
Time Frame: From ED arrival through Day 28
Population: Patients with at least at 2 day stay in the ICU
Measure: Number; unit: participants
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 24 | 35
participants | 3 | 8
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; percent difference = -10.4, 95% CI 2-sided [-29.6 to 8.8]

13. Secondary Outcome: Acute Renal Failure Classification Score of "Failure" Without Glomerular Filtration Rate (GFR)
Description: Increased plasma creatinine > 3 x reference measure (ED admission) or acute plasma creatinine = 350 umol/L or acute rise = 44 umol/L or urine output < 0.3 mL/k/h x 24h. Only measured for patients with at least 2 days of ICU stay assessed.
Time Frame: From ED arrival through the first 24 hours
Population: Patients with at least at 2 day stay in the ICU
Measure: Number; unit: participants
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 24 | 35
participants | 1 | 3
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; percent difference = -4.4, 95% CI 2-sided [-16.6 to 7.8]

14. Secondary Outcome: Ventilator Free Days Through Day 28
Description: The number of days beginning with the day of the 911 call counted as "Day 0" through Day 28 during which the patient did not require mechanical ventilation. Deaths are assigned the worst score (0).
Time Frame: From day of the 911 call through Day 28
Population: Patients with known discharge status.
Measure: Mean (Standard Deviation); unit: Ventilator-free days
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 91 | 95
Ventilator-free days | 23.6 (10.7) | 24.5 (9.5)
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.8 to 2.1]

15. Secondary Outcome: Days Alive Out of the Intensive Care Unit (ICU) Through Day 28
Description: The number of days beginning with the day of the 911 call counted as "Day 0" through Day 28 during which the patient is alive and not being cared for in the intensive care unit
Time Frame: From day of the 911 call through Day 28
Population: Patients with known discharge status
Measure: Mean (Standard Deviation); unit: ICU-free days
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 91 | 95
ICU-free days | 23.0 (10.7) | 23.6 (9.8)
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-3.6 to 2.4]

16. Secondary Outcome: Days Alive Out of the Hospital Through Day 28
Description: The number of days beginning with the day of the 911 call counted as "Day 0" through Day 28 during which the patient is alive and not being cared for in the hospital
Time Frame: From day of the 911 call through Day 28
Population: Patients with known discharge status
Measure: Mean (Standard Deviation); unit: Days alive out of hospital thru day 28
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 91 | 95
Days alive out of hospital thru day 28 | 18.6 (10.3) | 18.5 (10.5)
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-2.9 to 3.1]

17. Secondary Outcome: Blunt Trauma 24 Hour Mortality
Description: The 24 hour mortality endpoint for the total number of patients injured by blunt mechanisms in each arm.
Time Frame: From time of hospital arrival through first 24 hours
Population: Analyzed patients had traumatic shock due to blunt traumatic mechanisms. One patient randomized to the controlled resuscitation group was not analyzed because neither blunt force nor penetrating injury had occurred. It was determined that the source of bleeding was from a gastrointestinal lesion.
Measure: Number; unit: participants
Groups:
- Controlled Resuscitation: Patients in the CR group received a 250 milliliter (ml) bolus of saline only if their SBP was < 70 millimeters of mercury (mmHg) or they had no palpable radial pulse.
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation
Number analyzed (Participants) | 62 | 63
participants
  Died within first 24 hours after hospital arrival | 11 | 2
  Alive at 24 hours after hospital arrival | 51 | 61
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation; Test type: Superiority or Other; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.03 to 0.92] — Adjusted for age (linear spline with knot at 45 years) and Injury Severity Score (ISS). ISS multiply imputed for one patient

18. Secondary Outcome: Penetrating Trauma 24 Hour Mortality
Description: The 24 hour mortality endpoint for the total number of patients injured by penetrating mechanisms in each arm.
Time Frame: From time of hospital arrival through first 24 hours
Population: Patients with traumatic shock due to penetrating traumatic mechanisms
Measure: Number; unit: participants
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation
Number analyzed (Participants) | 33 | 32
participants
  Died within first 24 hours after hospital arrival | 3 | 3
  Alive at 24 hours after hospital arrival | 30 | 29
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation; Test type: Superiority or Other; Odds Ratio (OR) = 1.92, 95% CI 2-sided [0.19 to 19.11] — Adjusted for age (linear spline with knot at 45 years) and Injury Severity Score (ISS)

19. Secondary Outcome: In-hospital Mortality
Description: Number of patients who died prior to discharge.
Time Frame: From day of the 911 call through hospital discharge
Population: All enrolled patients
Measure: Number; unit: participants
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Number analyzed (Participants) | 91 | 95
participants | 15 | 8
Statistical Analysis 1: Comparison: Standard Resuscitation (SR) vs Controlled Resuscitation (CR); Test type: Superiority or Other; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.22 to 1.77] — Adjusted for age (linear spline with knot at 45 years), penetrating mechanism (yes/no), and ISS (linear)

ADVERSE EVENTS:
Time Frame: Data were collected from the time the blinded study fluid kit was opened by the paramedic prior to hospital arrival to discharge, an average hospital stay of 7.6 days (SD 13.2).
Description: One CR patient enrolled as prisoner, which prohibited study data collection.
Groups:
- Controlled Resuscitation (CR): Patients in the CR group received a 250 milliliter (ml) bolus of saline only if their SBP was < 70 millimeters of mercury (mmHg) or they had no palpable radial pulse.
  The total number of patients at risk is one less than the total number of patients enrolled. Regulatory restrictions for prisoners required that no data collection, including severe adverse events, be performed for the patient who was determined to have been in police custody at the time of enrollment.
Arm/Group | Standard Resuscitation (SR) | Controlled Resuscitation (CR)
Serious Adverse Events (participants affected / at risk) | 8/95 | 18/96
Other Adverse Events (participants affected / at risk) | 0/95 | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Resuscitation (SR) (N=95) | Controlled Resuscitation (CR) (N=96)
Pneumonia (Infections and infestations) | 2 (2) | 6 (6) — Documented in the discharge note. Collected during chart review.
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3) — Documented in the discharge note. Collected during chart review.
Wound infection (Infections and infestations) | 0 (0) | 5 (5) — Documented in the discharge note. Collected during chart review.
Sepsis (Infections and infestations) | 1 (1) | 1 (1) — Documented in the discharge note. Collected during chart review.
Bloodstream infection (Infections and infestations) | 0 (0) | 1 (1) — Documented in the discharge note. Collected during chart review.
Intra-abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) — Documented in the discharge note. Collected during chart review.
Renal impairment (Renal and urinary disorders) | 3 (3) | 7 (7) — Documented in the discharge note. Collected during chart review.
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) — Documented in the discharge note. Collected during chart review.
Deep vein thrombosis (DVT) (Vascular disorders) | 1 (1) | 2 (2) — Documented in the discharge note. Collected during chart review.
Pulmonary embolus (Vascular disorders) | 0 (0) | 1 (1) — Documented in the discharge note. Collected during chart review.
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) — Documented in the discharge note. Collected during chart review.

LIMITATIONS AND CAVEATS:
One patient was determined to have been in police custody at the time of enrollment, which was a protocol violation. This patient was randomized to the controlled resuscitation group but was not included in the primary or secondary outcome analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research activities of the Resuscitation Outcomes Consortium (ROC) are intended to contribute applicable knowledge to the field of Resuscitative Medicine. Definitive contributions are made through publications in peer-reviewed literature. No participating institution may present or publish individual findings from work performed on study protocols without approval of the Publications Subcommittee (PS).